CLINICAL TRIAL: NCT02476513
Title: Clinical and Molecular Assessment of Men With High Risk for Esophageal Disorders
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: UAB 1354
Record Dates: First submitted 2014-10-27; First posted 2015-06-19 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Esophageal Diseases
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The H&E sections of all biopsy specimens will be reviewed by a GI diagnostic pathologist, Leona Council, MD, for histopathologic parameters including histologic grade and type. The histology will be characterized according to the scale depicted in figure 1, where 0 represents the earliest possible injury and 3 represents malignancy. All specimens will be processed in the typical manner, but reviewed by Dr. Council in the pathology department.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this study,the investigators will evaluate participants that have clinical features associated with an increased risk of esophageal disorders.The investigators will also see if there is a positive association of esophageal disorders in men,40-60 with or without abdominal obesity in the diagnosis of the following diseases; Gastroesophageal reflux disease, Barrett Esophagus and Esophageal Adenocarcinoma. The investigators hypothesize that most obese patients referred for Esophagogastroduodenoscopy will exhibit esophageal disorders. Since currently the rates of obesity and adenocarcinoma of the esophagus have increased significantly over the past 15 years, the investigators hope to find biochemical markers (i.e. pro-inflammatory mediators) in the esophagus. The investigators hope these samples will lead us to a differential expression of molecular markers and inflammatory mediators in the varying degrees of esophageal disorder

DETAILED DESCRIPTION:
Patients with elevated central adiposity have an increased risk of esophageal disorders; we will correlate central adiposity with advanced esophageal pathologies (BE and EAC). This will be done by comparing body mass and fat distribution to tissue abnormalities found by pathology review of EGD biopsy. It is anticipated that the group of men in this study will have an increased likelihood of histopathologic alteration, which we will fit into our scale (0-no inflammation, 1-inflammation or BE, 2-BE with dysplasia, and 3-carcinoma) according to the referral pattern at UAB's outpatient gastroenterology clinic.

At the molecular level, there is also a relationship between pro-inflammatory cytokines and obesity, which may contribute to esophageal disorder [28]. Metabolically active fat cells secrete cytokines exclusive to adipose tissue (adipokines, leptin/adiponectin) as well as the more classic signaling molecules, tumor necrosis factor alpha (TNF-α); interleukins (IL)-1, IL-6, IL-8, and IL-10; monocyte chemoattractant protein 1 (MCP-1); and macrophage inflammatory protein 1 (MIP 1) [29-33]. Obesity-triggered pro-inflammatory molecules may promote tissue injury, leading to metaplasia and dysplasia in BE and, subsequently, to carcinoma.

Thus, by measuring these pro-inflammatory markers in our prospective patient population, it will be determined if patients with elevated levels exhibit pathologic disorders in the esophagus and if the differential expression of these molecular markers correlates with degree of esophageal disorder. We will analyze samples collected from men for adipocytokines and for inflammatory mediators that are released with tissue injury. Additionally, we will examine molecular markers that correlate with more advanced esophageal disorders (BE with high grade dysplasia and EAC).

Persistent stimulation is needed to cause stepwise progression from the early stages of esophageal injury, to BE, to carcinoma. Since the molecular events that lead to this transformation are not known, our goal is to profile biopsy tissues collected from the prospective cohort of 60 men, analyzed by IHC for p53, Ki67, cyclin D1, IL-6, IL-8, Cox-2, DKK-1, CD44, leptin, and adiponectin. These molecules are known to be involved in transformation of normal esophageal epithelium to EACs via progression from metaplasia and BE to low-grade dysplasia and high-grade dysplasia. [34]. The clinical outcome measurements will be correlated with the levels of these molecules, determined by IHC, with metaplasia, degree of dysplasia in BE, and stage of EAC. For BE tissues, there is a correlation between the extent of p53 staining and aggressive clinical features. Our preliminary findings on six BEs, selected from the patient population at UAB, indicate that a high proportion of p53 staining directly correlates with high-grade lesions

ELIGIBILITY:
Inclusion Criteria:

1. Men only who are referred for upper endoscopy for the first time.Or who have had normal upper endoscopy in the last 10 years
2. Age criteria: 25-75 years in age
3. Patients undergoing EGD and willing to also consent to tissue biopsy, blood work and CT scan.
4. ECOG PFS 0-1

Exclusion Criteria:

1. Unstable medical condition, such as uncontrolled diabetes mellitus or hypertension or active infections requiring systemic therapy
2. Clinical evidence of cardiac or pulmonary dysfunction including, but not limited to, unstable congestive heart failure, uncontrolled arrhythmias, unstable coagulation disorders, or recent myocardial infarction (within 6 months)
3. Documented history of erosive esophagitis or non-erosive esophageal luminal. No prior history of Barrett's esophagus.

Ages: 25 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The goal of the study is to further clarify the relationship among esophageal disorders, obesity and inflammatory mediators that may identify a high risk patient profile that would warrant more frequent screening. We will accrue 60 men between the ages of 25 and 75 who are referred for upper endoscopy for the first time or subject who have had a normal upper endoscopy in the last 10 years. It is anticipated that some of the participants will not have symptoms of reflux or dyspepsia. Due to the pattern of referral, however, most will exhibit risk factors of esophageal disorders.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Correlation of obesity and increase risk of esophageal adenocarcinomas | 1-2 years
  We will use data collected from the waist measurements and the measurement compiled from the CT scan of the abdomen. The correlate it with the actual tissue markers(if any) found from the pathologists review.

SECONDARY OUTCOMES:
Developing a group of tissue markers that specifically relates to a increase in esophageal cancer | 1-2 years
  The pathologist and bio-marker laboratory will use the blood samples and tissue to provide a assay that can be used later to provide insight into the increase risk of developing Barrett's esophagus or esophageal adenocarcinoma

CONTACTS AND LOCATIONS:
Overall Officials: James A Posey, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States